CLINICAL TRIAL: NCT07277686
Title: AI Facial Analysis Algorithm to Screening Coronary Artery Disease in High-Risk Community Population
Status: Recruiting | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Collaborators: Zhoukou Specialized Disease Hospital (Unknown); Zhoukou Chuanhui District Hospital of Traditional Chinese Medicine (Unknown); Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Zhoukou Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-ZX165
Record Dates: First submitted 2025-11-29; First posted 2025-12-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease (CAD); Artificial Intelligence Algorithms; Face; Screening
MeSH Terms: conditions — Coronary Artery Disease; Facies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Diagnostic Test Cohort: Participants in this cohort undergo facial image-based AI screening. Subsequently, all participants in this group will undergo Coronary Computed Tomography Angiography (CCTA) as the gold standard reference to verify the diagnosis of CAD. All participants are followed up for 6 months.
  Interventions: Other: No Intervention
- Real-world Observational Cohort: Participants in this cohort represent a real-world setting. They are followed up for 6 months to observe the natural detection rate of CAD and the occurrence of MACE outcomes.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — No Intervention

SUMMARY:
This study aims to evaluate the effectiveness of this facial image-based AI algorithm for screening CAD in high-risk community populations (specifically individuals with diabetes, hypertension, or aged over 65). The main objectives are:

1. To verify if the AI algorithm can accurately distinguish between high-risk and low-risk groups by comparing the actual prevalence of CAD in these groups.
2. To compare the CAD detection rate using this AI screening strategy against the natural detection rate in a real-world cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years.
* Community high-risk population, defined as individuals meeting at least one of the following criteria:

  1. Diagnosed with Diabetes Mellitus;
  2. Diagnosed with Hypertension;
  3. Advanced age (> 65 years old).

Exclusion Criteria:

* Prior confirmed diagnosis of Coronary Heart Disease (CAD), including clinically diagnosed CAD, history of Coronary Artery Bypass Grafting (CABG), or history of Percutaneous Coronary Intervention (PCI).
* History of diagnosed Heart Failure.
* Significant facial alterations or conditions that may interfere with AI image analysis, such as plastic surgery, severe facial trauma, or heavy makeup.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of community-dwelling residents identified as high-risk for Coronary Heart Disease (CHD). Participants are recruited from local community health centers and primary care settings. The cohort primarily comprises elderly individuals (aged > 65 years) and those with established cardiovascular risk factors, specifically diabetes mellitus and hypertension, who have not been previously diagnosed with CHD.
Sampling Method: Non-Probability Sample
Enrollment: 1392 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Difference in Prevalence of CAD Between AI-Stratified High-Risk and Low-Risk Groups | Up to 6 months
  Participants in the diagnostic test cohort are stratified into high-risk and low-risk groups using the AI screening strategy. Subsequently, all participants undergo Coronary Computed Tomography Angiography (CCTA). This outcome measures the difference in CAD prevalence between the two groups based on CCTA results.

SECONDARY OUTCOMES:
The detection rate of CAD | 6 months
  The detection rate of CAD
Incidence of Major Adverse Cardiovascular Events (MACE) | 6 months
  MACE is defined as a composite endpoint including all-cause death, myocardial infarction, and ischemia-driven coronary revascularization. The incidence of MACE will be compared between the diagnostic test cohort and the real-world observational cohort.
Incidence of All-Cause Death | 6 months
  The number of participants who die from any cause during the follow-up period.
Incidence of Myocardial Infarction | 6 months
  The number of participants who experience a myocardial infarction event, diagnosed based on standard clinical guidelines (e.g., symptoms, ECG changes, and troponin elevation).
Incidence of Ischemia-Driven Coronary Revascularization | 6 months
  Defined as any percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) driven by ischemic symptoms or objective evidence of ischemia.
Incidence of Screening-Driven Coronary Revascularization | 6 months
  Defined as coronary revascularization procedures (PCI or CABG) triggered by findings from screening examinations rather than acute clinical symptoms.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Zhoukou Chuanhui District Hospital of Traditional Chinese Medicine, Zhoukou, Henan
  - Zhoukou Specialized Disease Hospital, Zhoukou, Henan
  - Fuwai Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing

IPD SHARING:
Plan to Share IPD: No